CLINICAL TRIAL: NCT06350136
Title: The Effect of Self-Management Support Provided to Hypertension Patients Affected by the Earthquake Via Tele-Nursing on Patients' Treatment Compliance and Self-Care Management: A Randomized Controlled Study
Brief Title: The Effect of Self-Management Support Provided to Hypertension Patients Affected by the Earthquake Via Tele-Nursing on Patients' Treatment Compliance and Self-Care Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Gülcan Bahçecioğlu Turan, Principal Investigator, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/05-37
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: With Tele-Nursing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With Tele-Nursing (Experimental): With Tele-Nursing
  Interventions: Behavioral: With Tele-Nursing
- Control (No Intervention): no With Tele-Nursing

INTERVENTIONS:
Behavioral: With Tele-Nursing — no With Tele-Nursing
  Other Names: Control
  Arms: With Tele-Nursing

SUMMARY:
This important research includes a randomized controlled trial evaluating the potential of self-management support provided via telenursing to earthquake-affected hypertension patients to improve patients' treatment adherence and overall self-care management. This study will be carried out at Fırat University Hospital and will cover a wide range of effects on health outcomes in individuals receiving hypertension treatment. The sample selected from hypertension patients, which constitute the population of the research, was based on predetermined power analysis criteria. It has been determined that at least 51 hypertension patients should be included in each of the intervention and control groups, and accordingly, a total of 150 hypertension patients will be included in the study.

. The results obtained within this framework may provide guidance in the development and implementation of Turkey's health policies, and may also shed light on strategies for the management of other similar health problems. On the other hand, strengthening the digital health infrastructure and effective management of chronic diseases, which are among the health-related targets of the Development Plan, further emphasize the importance of this research. The success of the self-management model supported by tele-nursing can serve as an example in the integration of digital health technologies into Turkey's healthcare system and be an important step towards achieving strategic goals in this field.

ELIGIBILITY:
Inclusion Criteria:

* Being followed for at least 6 months with the diagnosis of essential hypertension,

  * Patients diagnosed with hypertension who suffered financial or moral loss after the earthquake
  * Located in Elazığ at the time of the February 6 earthquake
  * Continuing to live in Elazığ after the earthquake
  * Using antihypertensive medication,
  * No change in antihypertensive drug treatment has been made in the last month,
  * Computer/tablet/smartphone etc. to watch videos. having technological devices,
  * Having internet access,
  * Being over 40 years old,
  * Education level must be at least primary education level

Exclusion Criteria:

* Being pregnant or breastfeeding
* Presence of another accompanying chronic disease (Diabetes mellitus, cancer, chronic renal failure, chronic obstructive pulmonary disease, heart failure, etc.),
* Having physical (speech, hearing impairment, etc.), neurological and psychological problems that prevent filling out research forms and participating in training.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Hill-Bone Hypertension Treatment Compliance Scale | 12 week
  The scale consists of 14 questions. On a four-point Likert scale (0=never, 1=sometimes, 2=most of the time and 3=always), interview (items 6, 7 and 8), medical (items 1, 2, 9, 10, 11, 12, 13) and 14) and nutrition (items 3, 4 and 5). Except for the 6th question of the scale, all other questions are in the form of negative questions. Total scores from the scale vary between 0 and 42, with 0 points indicating perfect compliance with treatment. A high total score from the scale indicates decreased compliance with treatment.
Self-Care Management Scale in Chronic Diseases; | 12 week
  The scale consists of 35 items and is a five-point Likert type (1=strongly disagree, 2=disagree, 3=undecided, 4=agree, 5=strongly agree). The scale includes self-protection (items 2, 6, 8, 11, 15, 18, 19, 20, 22, 23, 25-34), and social protection (items 1, 3, 4, 5, 7, 9, 10, 12). It has two sub-dimensions: , 13, 14, 16, 17, 21, 24 and 35 items). The 3rd, 15th, 19th and 28th items in the scale are negative statements. The total scores that can be obtained from the scale vary between 35-175 points, and an increase in the score indicates that the individual's self-care management also increases.
Psychological Impact of Earthquake Scale: | 12 week
  The scale consists of 41 items. The scale is a 5-point Likert (1: Strongly Disagree, 2: Disagree, 3: Neither Agree nor Disagree, 4: Agree, 5: Strongly Agree). There are 6 sub-dimensions. As the score on the scale increases, the psychological impact of the earthquake on individuals increases. Scale Cronbach's Alpha values vary between 0.84 and 0.96.
Earthquake Stress Coping Strategies Scale | 12 week
  The scale consists of 16 items and has 3 subscales. A 4-point rating was used in the scale: Always (4) and Never (1). However, in the Social Support Seeking subscale, Item 4 (I try to keep my feelings to myself) and Item 12 (I prefer not to talk about my fears and concerns) are scored in the opposite direction because they indicate that the individual does not seek social support. The score ranges of the Religious Coping and Social Support Seeking subscales, each consisting of 5 items, are 5-20, and the score range of the Positive Reappraisal subscale, consisting of 6 items, is 6-24. A high score for each dimension indicates that the individual uses that coping strategy more, while a low score indicates that the individual uses it less

IPD SHARING:
Plan to Share IPD: No